CLINICAL TRIAL: NCT06265467
Title: Assessment of Implants Placed Simultaneously With Maxillary Sinus Bone Augmentation Using Two Different Sinus Elevation Techniques: A Randomized Control Clinical Trial
Brief Title: Evaluation of Two Different Techniques for Sinus Elevation, Open Versus Closed .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Collaborators: Suez Canal University (Other)
Responsible Party: Principal Investigator, Hebatallah Abdo's Elsaid Mattar, Assisstant Lecturer, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28909108800228
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Alveolar Ridge Augmentation; Sinus Floor Augmentation; Maxillary Sinus
Keywords: Dental Implant; Maxillary Sinus Augmentation; Sinus Elevation; Open Sinus Elevation; Closed Sinus Elevation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: it is a double blinded study, both the outcome assessor and statistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group- Closed Sinus elevation (Experimental): Maxillary sinus floor elevation using osteotomes through a crestal approach. Followed by bone grafting using allogenic bone graft and simultaneous dental implant placement.
  Interventions: Procedure: Closed Sinus Elevation
- Control Group- Open sinus elevation (Active Comparator): Maxillary sinus floor elevation using sinus elevation tools through a lateral window approach. Followed by bone grafting using allogenic bone graft and simultaneous dental implant placement.
  Interventions: Procedure: Open Sinus Elevation

INTERVENTIONS:
Procedure: Closed Sinus Elevation — using a unique design of osteotomes to crestally elevate the Schneiderian membrane of the maxillary sinus floor
  Other Names: Crestal approach to elevate the maxillary sinus membrane; Osteotome Technique
  Arms: Test Group- Closed Sinus elevation
Procedure: Open Sinus Elevation — using a unique design of sinus elevators to laterally elevate the Schneiderian membrane of the maxillary sinus floor
  Other Names: Lateral Approach to elevate the maxillary sinus Membrane
  Arms: Control Group- Open sinus elevation

SUMMARY:
A clinical Trial, comparing two different techniques to elevate the maxillary sinus floor membrane to allow for simultaneous dental implant placement in the severely atrophied maxillary ridges.Both using allogenic bone substitute as the bone graft material. One technique is the open lateral window technique and the second is the closed crestal technique.

DETAILED DESCRIPTION:
Following extraction of posterior teeth in the maxillary arch, maxillary sinus pneumatization may pause a difficulty for dental implant placement. This difficulty may be overcome by maxillary sinus elevation with or without bone grafting or the use of short implants. Yet the literature available does not give conclusive answers as to what is the best approach for each clinical situation.

Aim of this study is to evaluate implants placed simultaneously with maxillary sinus bone augmentation using two different sinus floor elevation techniques. Null Hypothesis: There is no statistically significant difference between implants placed with crestal sinus approach and lateral sinus floor elevation, using bone grafting in both techniques, regarding implant stability and radiographic bone height gain.

Alternative Hypothesis: There is statistically significant difference between implants placed with crestal sinus approach and lateral sinus floor elevation, using bone grafting in both techniques, regarding implant stability and radiographic bone height gain.

Thirty implants in patients having posterior edentulism with maxillary sinus pneumatization were studied. All patients were be randomly allocated into two groups, group 1 (test group) had dental implants placed after crestal approach for sinus elevation, while group 2 (control group) had dental implants placed after lateral approach for maxillary sinus elevation. Both groups received allogenic bone grafts in the elevated sites. To assess implant stability, a resonance frequency analysis (RFA) device was used, for each implant the implant stability quotient (ISQ) values was measured on four sites over the implant. Mean values were calculated for each implant from the four recorded values. ISQ values were recorded immediately post-implant insertion, 9 months (after delivery of the final prosthesis) and at 12 post- operative. Cone Beam Computed Tomography (CBCT)s were made at 6 and 12 months post-operative to evaluate the radiographic bone changes in vertical dimension of bone height gained around each implant.

Steps of the clinical Procedures:

1. Clinical and radiographic evaluation:

   1. Evaluation of the patient's general condition of the oral cavity, to make sure it complies with the criteria required to be enrolled in the study in terms of oral hygiene, pathological conditions, occlusion and inter-arch space.
   2. A preoperative CBCT was performed for each patient prior to the surgery. Evaluation of available bone height and bucco-palatal bone width. Suitable implant length and diameter will be determined as well.
2. Random allocation:

   The patients were divided into two groups with a random allocation sequence generator.
3. Surgical procedure:

   After administration of local anesthesia, the allocation was revealed, for the test group, a full thickness flap was elevated at the edentulous site with two vertical releasing incision and then the preparation of osteotomy was prepared following standard implant system protocol preparation of the osteotomy. Drilling was done gently till reaching 0-1mm from the sinus floor, then in fracture of the sinus floor was done using osteotomes followed by bone grafting to raise the sinus floor from 3-5 mm and finally implant placement. For the control group, a full-thickness flap was elevated at the edentulous site with two vertical releasing incisions extending to the vestibule for better reflection and exposure to the lateral wall of the sinus. The lateral antrostomy was prepared in the lateral sinus wall using rotary bur no. 8 to provide adequate access to remove the thin to thick cortical bone and to expose the thin sinus membrane. The membrane was elevated across the sinus floor and up the medial wall and this elevation extended anteriorly-posteriorly to provide the exposed sinus floor. Drilling was done gently till reaching 0-1mm from the sinus floor, then implant placement and bone grafting took place. Primary stability of the implant was measured by rotational insertion torque value, to be ≥30 Nano centimeter(25). A resorbable collagen membrane was placed over the window preparation in the lateral approach to prevent the flap tissue from entering inside the antrostomy and the influencing the osseointegration process. Primary closure of the flap was achieved.
4. Postoperative Care:

Appropriate postoperative care was given to the patients and proper medications prescribed to them.

Patient self-care instructions:

* Application of an ice pack to the treated area for the first 24 hours will be instructed.
* The patients will be instructed to gently brush the operated area after two weeks with a soft brush.
* In case of emergency; severe pain and bleeding, the patient will be presented to the clinic.
* Patients will be recalled after two weeks for suture removal and every month for supportive periodontal therapy and recording of outcome variables at six,nine and twelve months.

After 9 months of the implant placement, stage II will be performed, 2 weeks later, impressions will be taken as regular for the prosthetic crowns fabrication. All crowns will be temporary cemented to allow an easy access to the implant platform for the follow-up RFA measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have at least one missing posterior maxillary tooth with sound adjacent teeth.
2. Adults above the age of 18.
3. Bone height from 4mm to 7mm under the maxillary sinus assessed in CBCT.
4. Good oral hygiene.
5. Patient accepts to sign an informed consent.

Exclusion Criteria:

1. Smokers (more than 10 cigarettes per day).
2. Medically compromised patients.
3. Patients with active infection related at the site of implant/bone graft placement.
4. Patients with untreated active periodontal diseases.
5. Patients with parafunctional habits.
6. Acute or chronic sinusitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Implant Stability | immediate postoperative- 9 months- 12 months
  Resonance Frequency analysis (RFA) a Device Named "Ostell" Device for measuring RFA

SECONDARY OUTCOMES:
Radiographic bone gain | immediate post-operative- 6 months-12 months
  CBCT linear measurements using the ruler tool in the CBCT software to assess radiographic vertical bone height gain in millimeter in both techniques

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elsholkamy, Professor, Study Director — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No